CLINICAL TRIAL: NCT02646813
Title: A Comparison of Intraluminal and Extraluminal Placement of the Arndt Bronchial Blockers for Adult Thoracic Surgery
Brief Title: Comparison of Intra and Extraluminal Bronchial Blocker in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00035615
Record Dates: First submitted 2015-12-31; First posted 2016-01-06 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Operative, Non Cardiac, Thoracic Disease
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraluminal Placement (Active Comparator): These patients will have the Arndt endobronchial blocker placed within the endotracheal tube for lung isolation during their thoracic surgery. The observer will measure time required to place blocker correctly prior to surgery.
  Interventions: Procedure: Intraluminal Placement
- Extraluminal Placement (Experimental): These patients will have the Arndt endobronchial blocker placed outside of the endotracheal tube for lung isolation during their thoracic surgery. The investigator will measure the time required for placement.
  Interventions: Procedure: Extraluminal Placement

INTERVENTIONS:
Procedure: Intraluminal Placement — Pt. will have Arndt Endobronchial Blocker placed intraluminally
  Arms: Intraluminal Placement
Procedure: Extraluminal Placement — Pt. will have Arndt Endobronchial Blocker placed extraluminally
  Arms: Extraluminal Placement

SUMMARY:
The objective of this study is to evaluate the time and ease of placement of an extra-luminal Arndt bronchial blocker versus placing it intra-luminally.

An additional objective will be to assess if there are any other significant clinical differences between these two approaches to placement of the BB including overall quality of isolation, an increase in post-operatives sore throat, post-operative hoarseness, and increased incidence of needing to reposition the blocker

DETAILED DESCRIPTION:
Once the patient is recruited in the preoperative assessment clinic, this information will be relayed to the study investigators. On the day of surgery the patient will then be randomized using a random number generator and opaque envelope method for group allocation to either intra-luminal or extra-luminal placement of a bronchial blocker.

The investigators will record age, height, weight, gender, American Society of Anesthesia Classification, type of surgery, sided of surgery, duration of surgery, duration, and anesthesia.

An IV will be placed in the patient prior to going to the OR. Once in the OR the patient will have routine monitors placed. The patient will be pre-oxygenated with 100% O2 for 2 minutes and induced with Propofol and rocuronium 0.8 mg/kg. The patient will then be hand ventilated with 100% oxygen. 3 minutes after administration of rocuronium the patient will have direct laryngoscopy performed with by one of the cardiac anesthesia fellows who has practiced placement of the BB both intraluminally and extraluminally in the simulator 10 times for each technique.

In the intra-luminal group the patient will be intubated with a 8.0 cuffed endotracheal tube(ETT). We will confirm endotracheal placement of the ETT via auscultation and ETCO2. The ETT will be secured at an appropriated depth, the blocker, y-piece, and flexible fiberoptic bronchoscope(FFB) set up will be assembled and placed onto the ETT in standard fashion recommended by the manufacturer for placement of an intra-luminal blocker. The fiberscope will then be advanced into the desired bronchus depending on the laterality of surgery. Once in place, the cuff will be inflated and isolation will be checked with auscultation. Time for initial bronchial blocker placement will be recorded from the point of the direct laryngoscopy(DL) to removal of the fiberscope after visualization of the bronchial blocker(BB) with the cuff inflated in the correct position.

In the extra-luminal group the patient will have the 9 Fr BB placed into the glottis and advanced to a depth of approximately 25 cm. Prior to placement, the blocker will be bent to roughly 45 degrees 2 cm proximal to the cuff balloon to facilitate placement of the blocker. The patient will then be intubated with an 8.0 cuffed ETT. We will confirm endotracheal placement of the ETT via auscultation and ETCO2. The ETT cuff should not be inflated to assure smooth movement of the blocker.

At this point a FFB will be introduced into the ETT to evaluate the position of the blocker. If the blocker is located in the correct mainstem bronchus the depth will be adjusted under direct vision. If it is not located on the correct side, the blocker will be withdrawn into the trachea and using a twisting motion will be manipulated and directed into the other side. Once in position the ETT cuff will be inflated. The BB cuff will be inflated and isolation will be checked with auscultation. Time for initial bronchial blocker placement will be recorded from the point of the DL to removal of the fiberscope after visualization of the BB with the cuff inflated in the correct position.

Other intravascular lines such as a radial arterial line and additional peripheral IV may be placed at the discretion of the attending anesthesiologist.

Following BB and line placement in both patient groups, the patient will be placed in the lateral position with the operative side up. Once in the final position prior to prepping and draping the blocker in both groups will be checked to make sure it is still correctly placed with a FFB. The blocker will be inflated under direct visualization and the patient will be placed on 100% O2.

The patient will be prepped and draped. The wire loop will be left in place in all patients in case the blocker needs to be repositioned until the end of the procedure. The lung will be allowed to passively deflate.

The surgeon will be queried as to the quality of isolation upon entry into the chest and this will be recorded. This will be based on a three point scale. Excellent, Fair, or Poor. This will be queried every 30 minutes for the duration of the procedure.

We will record any episodes of loss of isolation and details of repositioning including times and the issue of malposition i.e. the blocker slipped out or slipped in too far or suddenly slipped into the other mainstem bronchus. We will record any episodes of ongoing desaturation which require the deflation of the BB cuff and ventilation of both lungs.

At the conclusion of the intrathoracic portion of the procedure the BB cuff will be deflated and the lung on the operative side will be reinflated. The wire will be removed from the BB in both groups and the BB will be removed from the ETT in the intra-luminal group and the trachea in the extra-luminal group.

The patient will be extubated according to normal clinical practices and will be taken to the post anesthesia care unit.

The patient will be contacted on post-operative days 1 and 2 to assess for hoarseness and sore throat. The investigator will also record any significant morbidity or mortality events such as prolonged mechanical ventilation or cardiac arrest or stroke that may occur within the first 2 post-operative days.

The study will be performed at Wake Forest Baptist Medical Center a tertiary academic medical center.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and <80
* Patients scheduled for non cardiac, thoracic surgery requiring lung isolation

Exclusion Criteria:

* History of difficult airway/intubation
* Patients suspected to have a difficult airway
* Morbid obesity BMI >39
* Pregnancy
* Emergency status of surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time for placement of an extra-luminal Arndt bronchial blocker versus placing it intra-luminally | <8 minutes

SECONDARY OUTCOMES:
Sore Throat | <48hrs postop
  The investigator will query the study participants on post op days 1 and 2, and will use a qualitative scale from 1-4. 1-No Sore throat, 2-mild sorethroat, 3-moderate sorethroat, 4-severe sorethroat. The investigators will the compare means from the arms of the study.

OTHER OUTCOMES:
Quality of Lung Isolation | Duration of surgery
  The investigators will use a qualitative scale. 1-Perfect lung isolation and operative conditions. 2-Acceptable lung isolation and operative conditions, 3-No lung isolation and poor operative conditions. The surgeon will be queried every 30 minutes. The means for the two groups will be compared for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Templeton, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clayton-Smith A, Bennett K, Alston RP, Adams G, Brown G, Hawthorne T, Hu M, Sinclair A, Tan J. A Comparison of the Efficacy and Adverse Effects of Double-Lumen Endobronchial Tubes and Bronchial Blockers in Thoracic Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Cardiothorac Vasc Anesth. 2015 Aug;29(4):955-66. doi: 10.1053/j.jvca.2014.11.017. Epub 2014 Dec 2. PMID 25753765
- [Background] Campos JH, Hallam EA, Van Natta T, Kernstine KH. Devices for lung isolation used by anesthesiologists with limited thoracic experience: comparison of double-lumen endotracheal tube, Univent torque control blocker, and Arndt wire-guided endobronchial blocker. Anesthesiology. 2006 Feb;104(2):261-6, discussion 5A. doi: 10.1097/00000542-200602000-00010. PMID 16436844
- [Background] Knoll H, Ziegeler S, Schreiber JU, Buchinger H, Bialas P, Semyonov K, Graeter T, Mencke T. Airway injuries after one-lung ventilation: a comparison between double-lumen tube and endobronchial blocker: a randomized, prospective, controlled trial. Anesthesiology. 2006 Sep;105(3):471-7. doi: 10.1097/00000542-200609000-00009. PMID 16931978
- [Background] Hsieh VC, Thompson DR, Haberkern CM. Pediatric endobronchial blockers in infants: a refinement in technique. Paediatr Anaesth. 2015 Apr;25(4):438-9. doi: 10.1111/pan.12568. No abstract available. PMID 25752792
- [Background] Stephenson LL, Seefelder C. Routine extraluminal use of the 5F Arndt Endobronchial Blocker for one-lung ventilation in children up to 24 months of age. J Cardiothorac Vasc Anesth. 2011 Aug;25(4):683-6. doi: 10.1053/j.jvca.2010.04.020. Epub 2010 Jul 18. No abstract available. PMID 20638871
- [Background] Bastien JL, O'Brien JG, Frantz FW. Extraluminal use of the Arndt pediatric endobronchial blocker in an infant: a case report. Can J Anaesth. 2006 Feb;53(2):159-61. doi: 10.1007/BF03021821. PMID 16434756